CLINICAL TRIAL: NCT02340273
Title: Long Duration Therapeutic Ultrasound on Tendon Injuries
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: ZetrOZ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TN-02 (ZetrOZ-20140923)
Record Dates: First submitted 2015-01-12; First posted 2015-01-16 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Tendon Injuries; Musculoskeletal Pain
Keywords: tendinopathy; ultrasound; pain; heat; strength; LITUS; long duration; therapeutic ultrasound; tendonopathy
MeSH Terms: conditions — Tendon Injuries; Musculoskeletal Pain; Tendinopathy; Pain | interventions — Ultrasonic Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic ultrasound device (Experimental): Patients receive treatment from the long duration therapeutic ultrasound device for 4 hours every day for 6 weeks. The active device emits continuous ultrasound at 3 megahertz (MHz) frequency and 0.132 watts/cm2 intensity.
  Interventions: Device: Therapeutic ultrasound
- Placebo therapeutic ultrasound device (Placebo Comparator): Patients receive the "sham" long duration therapeutic ultrasound device for 4 hours every day for 6 weeks. The placebo device appears and operates identically to the active device except that it does not emit ultrasound.
  Interventions: Device: Placebo therapeutic ultrasound

INTERVENTIONS:
Device: Therapeutic ultrasound — Patients receive therapeutic ultrasound daily for 4 hours of continuous therapy at 3 megahertz (MHz) frequency and 0.132 Watts/cm2.
  Other Names: Therapeutic ultrasound (active); wearable ultrasound device; long duration ultrasound; LITUS device; long duration low intensity device
  Arms: Therapeutic ultrasound device
Device: Placebo therapeutic ultrasound — Patients receive "sham" therapeutic ultrasound daily for 4 hours.
  Arms: Placebo therapeutic ultrasound device

SUMMARY:
Human clinical trial to measure the effect of long duration therapeutic ultrasound on tendon injuries. The hypothesis is that use of long duration ultrasound will relieve pain, increase tendon strength, and improve quality of life for patients with tendon injury.

DETAILED DESCRIPTION:
The ability of long duration therapeutic ultrasound to reduce pain, increase strength, and improve quality of life for patients with tendon injury [e.g. tendinopathy of the elbow (medial or lateral], Achilles tendon, or patellar tendon) will be assessed. During the 7-week protocol, participants will receive 4 continuous hours of therapy daily.

For the first week, baseline data will be collected as participants report pain scores (VAS) in the morning, noon, and night. During the next 6 weeks, participants will self-apply the device each day and record their pain score (VAS) before and treatment; and record their pain score (VAS) while performing specified movements designed to evaluate tendon rehabilitation. At bi-weekly site visits, strength measurements will be performed on the injured and uninjured limb. Participants will also complete a standardized questionnaire to assess disability due to the specific tendon injury at baseline and study conclusion.

ELIGIBILITY:
Inclusion Criteria:

* Has been diagnosed with tendinitis in the elbow (medial or lateral epicondyles), patella, or Achilles tendon based on physical examination by a healthcare practitioner and medical history. Physical examination must include one of the following: assessment of pain during manual movements of the injured limb (e.g. a positive Mill's Test [Wadsworth, 1987] for elbow tendinitis), or local tenderness upon palpation over the tendon
* Experience tendon pain greater than 1 (using the VAS scale of 0-10) during the week preceding study screening
* Between 18 and 70 years of age
* Willing and able to self-administer the study device to the treatment area daily
* Have access to a mobile phone or camera to take a picture of the treatment area immediately after use of the device
* Body Mass Index (BMI) is less than or equal to 34.0
* Agree to document all pain medications and associated dosages during participation in the study.
* If taking prescription pain medication, agree to keep dosage constant (unchanged) during participation in the study.
* Agree not to use any topical solution such as analgesic cream or ointment on the treatment area during participation in the study

Exclusion Criteria:

* Subjects that cannot speak, read or write English
* History or current diagnosis of tendinosis or a tendon tear
* Known neuropathy (nerve damage that affects the treatment area)
* Surgery in the treatment area within the last 6 months
* Non-ambulatory (unable to walk)
* Prisoner
* Pregnant
* Have a pacemaker
* Malignancy in the treatment area
* Refuse to discontinue all other interventional treatment modalities (i.e. transcutaneous electrical nerve stimulation (TENS), electrical stimulation, or other ultrasound therapy) during the study
* Local corticosteroid or platelet-rich plasma (PRP) injection within the past 3 months
* Clinically significant or unstable medical or psychological conditions that would compromise participation in the study
* Participated in a clinical trial for an investigational drug and/or agent within 30 days prior to screening
* Involved in any injury-related litigation in the treatment area
* Open sores or wounds in the treatment area that would prevent use of the device
* Arthritis in the treatment area
* Carpal tunnel syndrome (if subject has elbow tendinitis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in pain on the visual analog scale (VAS) from baseline to study conclusion | Baseline, Week 7

SECONDARY OUTCOMES:
Pressure point sensitivity as measured through algometry | Baseline, Week 7
Change in pain during functional testing as measured by VAS | Baseline, Week 7
Change in strength of limb through dynamometry | Baseline, Week 7
Quality of life and functioning through limb-specific standardized questionnaires | Baseline, Week 7

CONTACTS AND LOCATIONS:
Overall Officials: George K Lewis, PhD, Principal Investigator — Sponsor GmbH
Locations (2):
- United States (2):
  - Clinical Research Consulting, Milford, Connecticut
  - Zetroz, Inc, Trumbull, Connecticut